CLINICAL TRIAL: NCT02465372
Title: Utilizing Physical Activity Coordinators to Increase Physical Activity Among Youth
Brief Title: Be a Champion! Comprehensive School Physical Activity Program
Acronym: BAC!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: University of South Carolina (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00038003; 1R21HL121692-01A1 (NIH)
Record Dates: First submitted 2015-05-21; First posted 2015-06-08 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: Motor Activity
Keywords: Physical Activity; Youth; School Health
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSPAP (Experimental): Schools in this arm will receive the Comprehensive School Physical Activity Program training.
  Interventions: Behavioral: CSPAP
- Control (No Intervention): Standard practice.

INTERVENTIONS:
Behavioral: CSPAP — Comprehensive School Physical Activity Program.
  Other Names: Be a Champion!
  Arms: CSPAP

SUMMARY:
The purpose of this project is to develop a Comprehensive School Physical Activity Program (CSPAP) training protocol, and test the feasibility, acceptability, and effectiveness of its delivery in an elementary school setting.

DETAILED DESCRIPTION:
Children across the United States are insufficiently physically active. In response, numerous physical activity (PA) interventions have been developed and tested, the majority within the school setting. Unfortunately, these have resulted in limited, if any impact on children's PA. The investigators feel that this absence of effect stems from a lack of tailoring at the school level and a resulting lack in institutionalization. To address the latter issue, the investigators feel that it is important to leverage existing resources and capitalize on existing policies. The state of South Carolina has instituted the role of "Physical Activity Coordinators" to promote PA among students across and beyond the school day. However, while these positions are mandated by state law, the individuals in these positions often lack the training and support to maximize their impact. Our long-term goal is to develop best practices to inform the national movement to train school PA Coordinators to deliver a Comprehensive School Physical Activity Program (CSPAP) within schools that can be disseminated across the country. The objectives of the current application are to: 1) modify and expand existing CSPAP training curricula for PA Coordinators; 2) deliver the enhanced PA Coordinator training in our pilot schools; 3) conduct process evaluation on the implementation of a CSPAP by the PA Coordinators, and 4) evaluate the effectiveness of the trainings to increase children's objectively measured PA. The goal of the proposed study is to determine the acceptability, feasibility, and effectiveness of properly train PA Coordinators to promote PA in elementary school children. This goal will be achieved through the following aims: AIM 1: Develop an enhanced CSPAP training course and resource toolkit for PA Coordinators. AIM 2: Determine the acceptability/feasibility of the enhanced PA coordinator training and the implementation of a Comprehensive School Physical Activity Program in an elementary school setting. AIM 3: Determine the effectiveness of trained PA coordinators to increase objectively measured PA in elementary school youth. the investigators will randomize four schools to receive the PA Coordinator training (n=2) or continue standard practice (n=2). A comprehensive process and impact evaluation will be conducted to determine acceptability of the intervention, factors influencing implementation fidelity/dose, and the effectiveness of the PA Coordinators to increase physical activity measured via accelerometry in children.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in grades 2 - 5 at the participating school sites.

Exclusion Criteria:

* Physical or mental impairment that would preclude physical activity or protocol compliance.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 599 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Moore, Ph.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Justin B. Moore, Columbia, South Carolina, United States

REFERENCES:
- [Derived] Singletary CR, Weaver G, Carson RL, Beets MW, Pate RR, Saunders RP, Peluso AG, Moore JB. Evaluation of a comprehensive school physical activity program: Be a Champion! Eval Program Plann. 2019 Aug;75:54-60. doi: 10.1016/j.evalprogplan.2019.04.003. Epub 2019 May 2. PMID 31102834

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Schools
Period: Overall Study
Arm/Group | CSPAP | Control
Started | 349; 3 Schools | 250; 2 Schools
Completed | 227; 3 Schools | 153; 2 Schools
Not Completed | 122; 0 Schools | 97; 0 Schools

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CSPAP | Control | Total
Number analyzed (Participants) | 227 | 153 | 380
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 227 | 153 | 380
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 75 | 202
  Male | 100 | 78 | 178

OUTCOME MEASURES:

1. Primary Outcome: Change in Youth Physical Activity
Description: Physical activity measured using an accelerometer at baseline and one-year follow-up (spring 2015 and spring 2016).
Time Frame: baseline and one-year follow-up
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | CSPAP | Control
Number analyzed (Participants) | 227 | 153
minutes/day
  baseline | 32.13 (16.91) | 36.47 (16.33)
  one-year follow-up | 33.16 (16.70) | 36.50 (16.69)

2. Secondary Outcome: Feasibility of the Be a Champion! Program
Description: Implementation monitoring to determine feasibility of the program as indicated by the percentage of planned tasks achieved with full fidelity and as determined by the number who, a) assembled an implementation team, b) completed all trainings, c) completed self-assessments, d) developed action plans, and e) executed at least one component of their action plans.
Time Frame: Up to nine months.
Measure: Number; unit: schools
Units Other Than Participants: Schools
Arm/Group | CSPAP | Control
Number analyzed (Participants) | 227 | 153
Number analyzed (Schools) | 3 | 2
schools | 3 | 2

3. Secondary Outcome: Acceptability of the Be a Champion! Program
Description: Number of schools that indicated BAC was acceptable, based upon qualitative and quantitative feedback from principals, classroom teachers, and implementation teams.
Time Frame: Up to nine months.
Measure: Number; unit: number of schools
Units Other Than Participants: Schools
Arm/Group | CSPAP | Control
Number analyzed (Participants) | 227 | 153
Number analyzed (Schools) | 3 | 2
number of schools | 3 | 2

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | CSPAP | Control
All-Cause Mortality (participants affected / at risk) | 0/227 | 0/153
Serious Adverse Events (participants affected / at risk) | 0/227 | 0/153
Other Adverse Events (participants affected / at risk) | 0/227 | 0/153

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes